CLINICAL TRIAL: NCT07204548
Title: Ivonescimab Consolidation After Concurrent/Sequential Chemoradiation for Unresectable Stage III NSCLC- A Phase II Study
Brief Title: The IVO-LUNG Study
Acronym: IVO Lung
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-236
Record Dates: First submitted 2025-09-02; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer (Stage III)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab as consolidation after definitive concurrent/sequential chemoradiotherapy (Experimental): Ivonescimab as consolidation after definitive concurrent/sequential chemoradiotherapy. Ivonescimab is given by 20mg/kg BW,q3w, last for one year.
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab is given after definitive concurrent/sequential chemoradiotherapy
  Other Names: AK112; AK-112

SUMMARY:
This Phase II, open-label, single-arm study evaluates the efficacy and safety of one-year Ivonescimab consolidation therapy in patients with unresectable Stage III NSCLC who have not progressed after definitive chemoradiotherapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, Phase II clinical study. The study plans to enroll previously untreated patients with Stage III (AJCC 8th edition) unresectable NSCLC who have not progressed after definitive concurrent/sequential chemoradiotherapy (≥2 cycles of platinum-based doublet chemotherapy). Induction therapy prior to concurrent or sequential chemoradiation is permitted. Subjects will receive Ivonescimab consolidation therapy for one year. The study aims to evaluate the efficacy and safety of Ivonescimab as consolidation therapy, alongside the exploration of efficacy-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntary written informed consent.
2. age: 18-75 years old
3. ECOG performance status: 0 or 1
4. With a life expectancy of ≥ 3 months.
5. Patients with radiologically confirmed, treatment-naïve, unresectable Stage III NSCLC (staged according to the American Joint Committee on Cancer, 8th edition) who did not progress after definitive concurrent/sequential chemoradiotherapy. Induction therapy prior to chemoradiotherapy was permitted.
6. Negative for EGFR L858R/19del, ALK fusion, ROS1 fusion, RET fusion, BRAF V600E mutation, NTRK fusion, and MET exon 14 skipping mutation.
7. Presence of at least one measurable lesion per RECIST v1.1, which is suitable for accurate and reproducible repeated measurements.
8. For the exploration of efficacy-related biomarkers, the submission of tumor tissue, peripheral blood, and stool samples is required. Patients with biologically unavailable samples may be granted an exemption from this requirement.
9. Adequate organ function based on examinations within 14 days prior to the initiation of study treatment.
10. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to the first dose (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test must be performed, and the serum result shall be considered definitive). If a female subject of childbearing potential engages in sexual activity with a non-sterilized male partner, the subject must use a highly effective method of contraception starting from screening and must agree to continue its use for 120 days after the last dose of the study drug; the decision to discontinue contraception after this time point should be discussed with the investigator.
11. Non-sterilized male subjects who engage in sexual activity with a female partner of childbearing potential must use a highly effective method of contraception from the start of screening until 120 days after the last dose; the decision to discontinue contraception after this time point should be discussed with the investigator.
12. The subject is willing and able to comply with scheduled visits, the treatment plan, laboratory tests, and other study requirements.

Exclusion Criteria:

1. Patients with non-small cell lung cancer (NSCLC) that contains a small cell carcinoma component.
2. History of other malignancies (except carcinoma in situ of the cervix, non-melanoma skin cancer, bladder carcinoma in situ, etc.) or presence of other life-threatening diseases that may affect the completion of the study.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study.
4. Imaging during the screening period shows tumor invasion or the presence of significant necrosis or cavitation, and the investigator judges that study entry would pose a bleeding risk.
5. History of severe bleeding tendency or coagulation dysfunction; presence of clinically significant bleeding symptoms within 1 month prior to the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or spitting up ≥1 teaspoon of fresh blood or small blood clots, or coughing up blood without sputum; subjects with blood-tinged sputum are allowed), epistaxis (excluding minor nosebleeds and blood-tinged postnasal drip); received continuous antiplatelet or anticoagulant therapy within 10 days prior to the first dose.
6. Tumor compression of surrounding vital organs (e.g., esophagus) accompanied by related symptoms, compression of the superior vena cava, or invasion of mediastinal great vessels, heart, etc.
7. Received non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for treating thrombocytopenia) within 2 weeks prior to the first dose; received Chinese herbal medicine or Chinese proprietary medicine with anti-tumor indications within 2 weeks prior to the first dose.
8. Previously received surgical resection and experienced postoperative recurrence of Stage III NSCLC.
9. History of non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoid therapy, or current non-infectious pneumonitis.
10. Presence of uncontrolled serous cavity effusion.
11. Presence of uncontrolled comorbid diseases, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements or impair the ability to provide written informed consent.
12. History of myocarditis, cardiomyopathy, or malignant arrhythmia. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or above), or vascular disease (e.g., aortic aneurysm at risk of rupture) requiring hospitalization within 12 months prior to the first dose, or other cardiac damage that may affect the evaluation of study drug safety (e.g., poorly controlled arrhythmia, myocardial ischemia); History of esophageal/gastric varices, severe ulcer, unhealed wound, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to the first dose; Any arterial thromboembolic event, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to the first dose; Acute exacerbation of chronic obstructive pulmonary disease within 1 month prior to the first dose; Current hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive medication.
13. Severe infection within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; Active infection requiring systemic anti-infective therapy within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C).
14. Active or history of definite autoimmune diseases, including but not limited to inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea), systemic lupus erythematosus, or other conditions unsuitable for treatment with immune checkpoint inhibitors.
15. History of immunodeficiency; Positive HIV antibody test; Current long-term use of systemic corticosteroids or other immunosuppressants.
16. Known active tuberculosis (TB); subjects suspected of having active TB require clinical evaluation to rule it out (e.g., sputum TB test, chest X-ray, etc.); Known active syphilis infection.
17. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
18. Subjects with active hepatitis B (HBsAg positive and HBV-DNA >1000 copies/ml or above the lower limit of detection); Subjects with active hepatitis C (HCV-RNA positive).
19. Major surgery or severe trauma within 30 days prior to the first dose, or planned major surgery within 30 days after the first dose (as determined by the investigator); Minor local surgery within 3 days prior to the first dose (excluding PICC line placement, port implantation).
20. Received live attenuated vaccines within 30 days prior to the first dose, or plans to receive live attenuated vaccines during the study period; Note: Live attenuated influenza vaccines cannot be administered within 90 days after the last dose of study treatment.
21. Known allergy to any component of the study drug; History of severe hypersensitivity reactions to other monoclonal antibodies.
22. Known history of mental illness, drug abuse, alcoholism, or substance abuse.
23. Pregnant or lactating women.
24. Any disease, treatment, or laboratory abnormality, historical or current, that may confound the study results, interfere with the subject's full participation in the study, or for which participation may not be in the best interest of the subject.
25. Uncontrolled metabolic disorders; or local or systemic diseases not caused by malignancy; or secondary diseases or symptoms caused by the tumor that could pose a high medical risk and/or uncertainty in survival evaluation, such as tumor-related leukemoid reaction (white blood cell count >20×10⁹/L), cachexia (e.g., known weight loss >10% in the 3 months prior to screening), etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
12-month PFS rate | From the date of enrollment untill 12 month
  The percentage of patients who has not experienced first documented progression or date of death from any cause, whichever came first, assessed up to 12 months from the date of enrollment.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | From the date of enrollment untill the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months"
  (Number of patients with CR + Number of patients with PR) / Total number of evaluable patients based on the RECIST V1.1
Progression free survival | From the date of enrollment to the date of first documented progression or date of death from any cause, assessed up to 100 months.
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
overall survival | From enrollment to death
  Survival time from enrollment to death
Treatment related adverse event | From enrollment to discontinuation of the study
  Any unfavorable and unintended sign, symptom, or disease that occurs in a participant during a clinical trial, which is deemed to have a reasonable possibility of being caused by the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Li-Kun Chen, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881